CLINICAL TRIAL: NCT02955693
Title: Randomized, Open-label, Single-center, Four-way Crossover, Single Dose Study to Investigate the Pharmacokinetics of LAS41008 120 mg Gastro-resistant Tablet and Fumaderm® 120 mg Gastro-resistant Tablet Under Fasting and Fed Conditions in Healthy Subjects
Brief Title: Study of the Effects of the Organism on Monomethyl Fumarate (MMF) After the Administration of LAS41008
Acronym: LAS41008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M-41008-08; PXL230623 (Other: PAREXEL International); 2016-002314-50 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-11-04 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Psoriasis
Keywords: Pharmacokinetics; Healthy volunteers; Monomethylfumarate; Dimethyl fumarate; Fumaderm®; Ethyl fumarate
MeSH Terms: conditions — Psoriasis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence A (n=8) (Other): Fumaderm® 120 mg fed (Period 1) - LAS41008 120 mg fasting (Period 2) -Fumaderm® 120 mg fasting (Period 3) - LAS41008 120 mg fed (Period 4)
  Interventions: Drug: LAS41008 120 mg / Fumaderm® 120 mg
- Sequence B (n=8) (Other): LAS41008 120 mg fasting (Period 1) - LAS41008 120 mg fed (Period 2) - Fumaderm® 120 mg fed (Period 3) - Fumaderm® 120 mg fasting (Period 4)
  Interventions: Drug: LAS41008 120 mg / Fumaderm® 120 mg
- Sequence C (n=8) (Other): Fumaderm® 120 mg fasting (Period 1) - Fumaderm® 120 mg fed (Period 2) - LAS41008 120 mg fed (Period 3) - LAS41008 120 mg fasting (Period 4)
  Interventions: Drug: LAS41008 120 mg / Fumaderm® 120 mg
- Sequence D (n=8) (Other): LAS41008 120 mg fed (Period 1) - Fumaderm® 120 mg fasting (Period 2) - LAS41008 120 mg fasting (Period 3) - Fumaderm® 120 mg fed (Period 4)
  Interventions: Drug: LAS41008 120 mg / Fumaderm® 120 mg

INTERVENTIONS:
Drug: LAS41008 120 mg / Fumaderm® 120 mg — Single dose of LAS41008 120 mg or Fumaderm® 120 mg in each Period
  Other Names: LAS41008: DMF / Fumaderm®: DMF + Ca, Mg and Zn salts of EHF

SUMMARY:
The purpose of this study is to determine how the organism affects MMF (metabolite of dimethyl fumarate [DMF]) after single oral dose administration of LAS41008 120 mg gastroresistant tablet and Fumaderm® 120 mg gastro-resistant tablet under fasting and fed conditions. The study also aims to assess the safety of the study treatments.

DETAILED DESCRIPTION:
The present study will be conducted to further investigate the pharmacokinetics (PK) of LAS41008 (containing DMF) after single oral dose administrations of a 120 mg gastro-resistant tablet under fed and fasting conditions.

Two previous Phase 1 studies allowed exploring the PK of LAS41008 30 mg and 120 mg separately after multiple dosing. In the current study, an improved bioanalytical method will allow the detection of lower MMF concentrations, and thus the same gastro-resistant tablet formulation (LAS41008) as used in the previous Phase 1 study will be investigated, but on a larger population and after single oral dose administration. Only the higher LAS41008 dose (120 mg) will be tested, as this is the formulation to be most frequently used during a standard treatment course for psoriasis with LAS41008. Similarly, single oral doses of Fumaderm® 120 mg (defined mixture of DMF and calcium (Ca), magnesium (Mg), and zinc (Zn) salts of ethylhydrogenfumarate (EHF, mono-ethyl fumarate (MEF)) will be tested in order to provide better comparative PK data. The comparison of LAS41008 and Fumaderm® PK will be evaluated in an exploratory manner.

The study will be conducted according to a randomised, open-label, four-way complete crossover, single dose design in 32 healthy male and female subjects. Up to 4 discontinued subjects may be replaced in case of early dropouts or a dropout rate greater than 15% (5 or more subjects). Gender balance will also be taken into consideration to ensure that roughly the same number of males and females are randomised. Upon inclusion into the treatment phase, each subject will be randomly allocated to one of four treatment sequences in a 4x4 Williams design. On Day 1 of each treatment period subjects will receive a single oral dose of either LAS41008 120 mg gastro-resistant tablet or Fumaderm® 120 mg gastro-resistant tablet under fasting or fed conditions. The drug administrations will be separated by a wash-out-phase of 7 ± 3 days. Blood sampling for PK will be performed until 24 hours after each study drug administration.

The Informed Consent Form (ICF) will be signed before any study activity, including the withdrawal of any concomitant medication (at least 2 weeks before this screening visit) if required for study participation. The Screening Visit will take place within 28 days before randomisation and after signing of the ICF to check subjects' eligibility. In each period, subjects will be admitted to the study centre from the morning of Day -1 until discharge in the morning of Day 2 (after collection of last blood sampling for PK).

The duration of study participation for each subject from Visit 1 (Screening) to the Follow-up Visit 7 ± 3 days after the last study drug administration is estimated to be approximately 7 to 10 weeks considering study visits time-window allowance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to understand and follow instructions during the study as determined by the Investigator.
* Signed and dated informed consent.
* Men and women of any ethnic origin between 18 and 55 years of age (inclusive, at the time of Screening) in general good physical health as determined by medical and surgical history, physical examination, ECG, vital signs, and clinical laboratory tests (including clinically significant changes in laboratory test).
* Weight within the normal range according to accepted values for the body mass index (BMI) within 18.0 to 29.0 kg/m2 (inclusive, at the time of Screening), and a body weight of at least 50 kg.
* Normal blood pressure (Systolic Blood Pressure ≥ 90, ≤ 139 mmHg; Diastolic Blood Pressure ≥ 55, ≤ 89 mmHg) measured after at least 5 minutes rest in supine position.
* A pulse rate of ≥ 45 and ≤ 99 beats per minute measured after at least 5 minutes rest in supine position.
* ECG recording, in triplicate, taken at least 1 minute apart; after at least 5 minutes of rest in a supine position without clinically significant abnormalities.

Exclusion Criteria:

* Subject who has received live-attenuated vaccine(s) within 4 weeks of Day 1 or plan to receive a vaccination during the study until 6 months after the last dose of study medication.
* More than moderate smoker (> 10 cigarettes/day).
* Demonstrating excess in xanthine consumption (more than five cups of coffee or equivalent per day).
* More than moderate alcohol consumption (subjects will be advised to consume no more than 2 units of alcohol per day and completely abstain from 72 hours prior to any visit (1 unit is equal to approximately 10 g of pure alcohol [250 mL] of beer [5%], 1 small glass [100 mL] of wine [12%] or 35 mL of spirits [35%]).
* Any history of alcohol or drug abuse or excessive intake of alcohol, as judged by the Investigator.
* Any history of drug hypersensitivity, asthma (with the exception of childhood asthma), urticaria or other severe allergic diathesis as well as active hay fever.
* Any history of hypersensitivity or lack of tolerability to the ingredients of the investigational medicinal product (IMP).
* Having febrile or infectious illness within at least 7 days prior to the Visit 1 (Screening) and Day -1 of Period 1.
* Any presence of acute or chronic liver or renal diseases.
* Any history or presence of gastrointestinal disease or problems including chronic gastritis, peptic ulcers, diarrhoea, or inflammatory bowel disease.
* Any history of clinically significant chronic or recurrent metabolic, pulmonary, neurological (especially history of epileptic seizures), endocrinological, immunological, psychiatric or cardiovascular disease, myopathies, and bleeding tendency.
* Subjects who have ever received immunosuppressant treatment (excluding topical or oral steroids taken 1 and 5 years before Visit 1 [Screening] respectively).
* Any history of frequent headache or migraine.
* Any history of malignancies (excluding basal skin cell cancer), as judged by the Investigator.
* Non-vasectomised man not using barrier contraception during the study.
* Nursing (breastfeeding) woman.
* Women with a positive serum pregnancy test at Visit 1 (Screening) or a positive urine pregnancy test on Day -1 of each Period or women of childbearing potential not using one highly effective method of birth control in combination with a barrier method during the study.
* Vegetarians.
* Unable or unwilling to comply with the dietary conditions in this study.
* Blood donation of more than 500 mL within 60 days prior to Visit 1 (Screening) or Day -1 of Period 1.
* Participation in the treatment phase of a clinical study within 90 days (or five half-life times, whichever is longer) prior to Visit 1 (Screening).
* Any abnormal safety laboratory values considered clinically significant by the Investigator, especially serum creatinine, alkaline phosphatase (AP), triglycerides or cholesterol, or medically relevant changes in haematology (especially differential cell count and thrombocytes), or relevant observations of protein in urine.
* Subjects with lymphocyte and white blood cell counts below the lower normal range (1.2 x 10^9L and 3.0 x 10^9L, respectively) or eosinophils above the upper normal range (0.4 x 10^9L) will not be included in the study.
* Liver enzyme results (aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT)) above the upper limit of normal (ULN female/male: AST: 31/37 IU/L; ALT: 35/50 IU/L; GGT: 42/71 IU/L).
* Creatinine values above the upper limit of normal and an estimated glomerular filtration rate below 90 mL/min.
* Positive test for human immunodeficiency virus (HIV) antibodies and antigen. Positive Hepatitis B virus surface antigen (HBsAg) test.
* Positive Anti-hepatitis C virus antibodies (Anti-HCV) test.
* Any history or suspicion of barbiturate, amphetamine, benzodiazepine, cocaine, opiates and cannabis abuse within the last 12 months (verified on-site by a urine test).
* Subject is not willing to refrain from xanthine-containing food or beverages as well as grapefruit products within 48 hour prior to first administration until discharge.
* Any gastrointestinal complaints within seven days prior to Visit 1 (Screening) or first study drug administration.
* Use of any medication (over the counter or prescription medication) within two weeks prior to Visit 1 (Screening) and Day -1 of Period 1 (or at least 10 times the respective elimination halflife, whichever is longer). Paracetamol may be concomitantly used, at the discretion of the Investigator (up to 1000 mg per day).
* Demonstrating any other active physical or mental disease, acute or chronic.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from zero to time t (AUC(0-t)) of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
  t is the time of the last concentration measured
Cmax of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
  Maximum plasma concentration
tmax of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
  Time to reach maximum plasma concentration
tlag of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
  Lag time

SECONDARY OUTCOMES:
Area under the concentration-time curve from zero to infinity (AUC) of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
Extrapolated part of AUC (%AUCext) of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
t1/2 of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
  Elimination half-life
Formation clearance of a drug to a metabolite (CL/f) of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
Vz/f of LAS41008 120 mg/Fumaderm® 120 mg | Within 1 hour pre-dose and post-dose at: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 13, 14, 16 and 24 hours (29 blood samples in each period)
  Apparent volume of distribution during terminal phase after non-intravenous administration

OTHER OUTCOMES:
Blood pressure | at Visit 1 (screening), 1 hour pre-dose and approximately at the same time on Day 2 of each period
Pulse rate | at Visit 1 (screening), 1 hour pre-dose and approximately at the same time on Day 2 of each period
Oral body temperature | at Visit 1 (screening) and pre-dose on Day 1 of each period
12-lead electrocardiogram (ECG) parameters | on Day 2 of each period
Physical examination findings | abbreviated on each admission and Day 2 of Period 4, and complete at Visit 1 (screening) and at the Follow-up Visit (7 ± 3 days after the study drug administration of the last treatment period)
Safety laboratory tests values (standard haematology, blood chemistry [clinical chemistry], urinalysis [sediment], and pregnancy test) | at Visit 1 (screening) and on Day 2 of each period, and at the Follow-Up Visit (7 ± 3 days after the study drug administration of the last treatment period)
  Note: Serum pregnancy test at Visit 1 (screening) and Follow-Up Visit; urine pregnancy test pre-dose
Overall tolerability (number of participants with adverse events (AEs) at the Follow-up Visit) | Follow-up Visit (7 ± 3 days after the study drug administration of the last treatment period)
Number of participants with adverse events/serious adverse events (SAEs) | from signature of the informed consent until the Follow-up Visit (7 ± 3 days after the study drug administration of the last treatment period)

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Godehard Ocker, MD, Study Director — Almirall Hermal GmbH
Locations (1):
- Almirall Investigational Site #1, London, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No